CLINICAL TRIAL: NCT06663059
Title: A Prospective, Multicenter, Exploratory Study Comparing 2 Cycles Versus 4 Cycles of Adebrelimab Combined With Chemotherapy as Neoadjuvant Treatment for Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Adebrelimab Neoadjuvant Treatment for Resectable ESCC: 2 vs 4 Cycles Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240709
Record Dates: First submitted 2024-08-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Squamous Cell Carcinoma; Adebrelimab; Neoadjuvant
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab combined with Chemotherapy 2 cycle (Experimental): Adebrelimab combined with albumin-bound paclitaxel and cisplatin for 2 cycles, followed by surgical resection.
  Interventions: Drug: Adebrelimab combined with albumin-bound paclitaxel and cisplatin 2 cycle
- Adebrelimab combined with Chemotherapy 4 cycle (Experimental): Adebrelimab combined with albumin-bound paclitaxel and cisplatin for 4 cycles, followed by surgical resection.
  Interventions: Drug: Adebrelimab combined with albumin-bound paclitaxel and cisplatin 4 cycle

INTERVENTIONS:
Drug: Adebrelimab combined with albumin-bound paclitaxel and cisplatin 2 cycle — Each treatment cycle is 3 weeks long (Q3W), with a total of 2 cycles. Adebrelimab: 1200 mg once on Day 1, administered intravenously, Q3W. Albumin-bound Paclitaxel: 130 mg/m² on Day 1 and Day 8, administered intravenously, Q3W.
  Cisplatin: 75 mg/m² on Day 1, administered intravenously, Q3W.
  Drug infusion should follow this sequence:
  Adebrelimab → Albumin-bound Paclitaxel → Cisplatin, with a minimum interval of 30 minutes between each infusion.
  Arms: Adebrelimab combined with Chemotherapy 2 cycle
Drug: Adebrelimab combined with albumin-bound paclitaxel and cisplatin 4 cycle — Each treatment cycle is 3 weeks long (Q3W), with a total of 4 cycles. Adebrelimab: 1200 mg once on Day 1, administered intravenously, Q3W. Albumin-bound Paclitaxel: 130 mg/m² on Day 1 and Day 8, administered intravenously, Q3W.
  Cisplatin: 75 mg/m² on Day 1, administered intravenously, Q3W.
  Drug infusion should follow this sequence:
  Adebrelimab → Albumin-bound Paclitaxel → Cisplatin, with a minimum interval of 30 minutes between each infusion.
  Arms: Adebrelimab combined with Chemotherapy 4 cycle

SUMMARY:
Observing the efficacy and safety of 2 cycles versus 4 cycles of Adebrelimab combined with chemotherapy as neoadjuvant treatment for patients with resectable locally advanced thoracic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, exploratory clinical trial. It involves patients with resectable locally advanced thoracic esophageal squamous cell carcinoma confirmed by histopathology or cytology. The study aims to compare the efficacy and safety of 2 cycles versus 4 cycles of Adebrelimab combined with chemotherapy as neoadjuvant treatment for these patients.

Eligible patients will be randomly assigned in a 1:1 ratio to either the 2-cycle group or the 4-cycle group. The primary endpoint is pathological complete response (pCR), with a planned enrollment of 80 patients.

The study consists of a screening period (from the signing of the informed consent form to the first administration of the drug, not exceeding 21 days), a treatment period (including neoadjuvant therapy and surgery), and a follow-up period (including safety follow-up, tumor progression/recurrence follow-up, and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed, and the participant must voluntarily join the study.
2. Histologically or cytologically confirmed esophageal squamous cell carcinoma.
3. Locally advanced thoracic esophageal cancer assessed by CT/MRI/EUS, with clinical staging T1b-4aN+M0 or T2-4N0M0 (T2N0 patients must have high-risk factors such as lymphovascular invasion [LVI], tumor size ≥3 cm, or poor differentiation) (according to AJCC 8th edition).
4. Expected to achieve R0 resection.
5. Age between 18 and 75 years, regardless of gender.
6. ECOG Performance Status 0-1.
7. No prior treatment for esophageal cancer, including radiotherapy, chemotherapy, or surgery.
8. Planning to undergo surgery after completing neoadjuvant therapy.
9. No contraindications for surgery.
10. Normal major organ functions, including:

    * **Hematology** (no use of blood components, growth factors, white blood cell stimulants, platelet stimulants, or anemia-correcting drugs within 14 days before the first use of the study drug):
    * Neutrophil count ≥1.5 × 10^9/L
    * Platelet count ≥100 × 10^9/L
    * Hemoglobin ≥90 g/L
    * **Biochemistry**:
    * Total bilirubin ≤1.5 × ULN
    * ALT ≤2.5 × ULN, AST ≤2.5 × ULN
    * Serum creatinine ≤1.5 × ULN, or creatinine clearance ≥50 mL/min
    * **Coagulation**:
    * International Normalized Ratio (INR) ≤1.5 × ULN
    * Activated Partial Thromboplastin Time (APTT) ≤1.5 × ULN
11. Female participants of childbearing potential must have a negative serum pregnancy test within 72 hours before starting the study drug and must use effective contraception (e.g., intrauterine device, contraceptive pills, or condoms) during the study and for at least 3 months after the last dose. Male participants with a fertile partner must be surgically sterilized or agree to use effective contraception during the study and for 3 months after the last dose.
12. Good compliance with the study and cooperation with follow-up.

Exclusion Criteria:

1. Tumor clearly invading adjacent organs (e.g., major arteries or trachea).
2. Supraclavicular lymph node metastasis.
3. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
4. Poor nutritional status, BMI < 18.5 kg/m²; if corrected with symptomatic nutritional support before randomization, may be considered for inclusion after assessment by the principal investigator.
5. History of allergy to monoclonal antibodies, Adebrelimab or its components, paclitaxel, cisplatin, or other platinum-based drugs.
6. Previous or current treatment with:

   * Any tumor-directed radiotherapy, chemotherapy, or other anti-tumor drugs.
   * Immunosuppressive drugs or systemic steroids (doses > 10 mg/day of prednisone or equivalent) within 2 weeks prior to the first use of the study drug; inhaled or topical steroids and adrenal corticosteroids for non-active autoimmune diseases are allowed.
   * Live attenuated vaccines within 4 weeks prior to the first use of the study drug.
   * Major surgery or severe trauma within 4 weeks prior to the first use of the study drug.
7. Active autoimmune diseases or a history of autoimmune diseases, including but not limited to: interstitial pneumonia, colitis, hepatitis, pituitaryitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (considered if on hormone replacement therapy); psoriasis or childhood asthma/allergy in complete remission without intervention can be considered, but those requiring bronchodilators for medical intervention cannot be included.
8. History of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiencies, or history of organ transplantation or allogeneic bone marrow transplantation.
9. Poorly controlled cardiac symptoms or diseases, including but not limited to: (1) NYHA Class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias not controlled or poorly controlled after clinical intervention.
10. Severe infection (CTCAE > 2) within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, or infection complications requiring hospitalization; active pulmonary inflammation on baseline chest imaging, symptoms and signs of infection within 14 days prior to the first use of the study drug, or need for antibiotic treatment, except for prophylactic use.
11. Active pulmonary tuberculosis infection discovered by medical history or CT, or history of active pulmonary tuberculosis within the past year, or history of active pulmonary tuberculosis more than 1 year ago without formal treatment.
12. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL) or hepatitis C (positive HCV antibody, and HCV RNA above the lower limit of detection).
13. Diagnosis of other malignant tumors within 5 years prior to the first use of the study drug, unless it is a low-risk malignancy (5-year survival rate > 90%), such as fully treated basal cell carcinoma, squamous cell skin cancer, or cervical carcinoma in situ.
14. Pregnant or breastfeeding women.
15. Any condition that, in the investigator's judgment, may lead to withdrawal from the study, such as other serious illnesses (including mental illnesses) requiring concurrent treatment, alcohol or drug abuse, family or social factors that may affect the participant's safety or compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate(pCR) | 7 days after surgery
  The lack of all signs of cancer in tissue samples removed during surgery or biopsy after treatment with radiation or chemotherapy.

SECONDARY OUTCOMES:
Major pathologic response (MPR) | 7 days after surgery
  MPR is defned as less than 10% residual viable tumor after neoadjuvant therapy.
R0 resection rate | postoperative 6 hours
  Proportion of R0 level surgery performed.
Event-free survival (EFS) | up to 2 years
  The length of time after primary treatment for a caancer ends that the patient remains free of certain complicationsor events that the treatment was intended toprevent or delay.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Dr, Study Chair — Tangdu hospital, The air force military university
Locations (1):
- Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No